CLINICAL TRIAL: NCT01943708
Title: A Study to Validate a Novel Auto Continuous Positive Airway Pressure Therapy
Brief Title: Novel Auto-continuous Positive Airway Pressure (CPAP) Validation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FPH-SA-10-07
Record Dates: First submitted 2011-07-10; First posted 2013-09-17 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous positive airway pressure (CPAP) device. (Active Comparator): Standard CPAP therapy
  Interventions: Device: CPAP
- Auto-CPAP device (SPAP). (Experimental): Novel Auto-CPAP algorithm
  Interventions: Device: SPAP

INTERVENTIONS:
Device: SPAP — Novel Auto-algorithm for Auto-CPAP device
  Arms: Auto-CPAP device (SPAP).
Device: CPAP — Standard CPAP therapy
  Arms: Continuous positive airway pressure (CPAP) device.

SUMMARY:
This single-blind randomised crossover trial aims to compare the efficacy of a novel Auto-CPAP algorithm (SPAP) to conventional CPAP. Up to 50 patients will be recruited from an OSA population, aged over 18.

DETAILED DESCRIPTION:
Auto-CPAP devices change therapeutic pressure based on the needs of the patient. Algorithms differ from machine to machine. This single-blind randomised crossover trial aims to compare the efficacy of SPAP (a novel Auto-CPAP algorithm) to conventional CPAP.

Up to 50 patients will be recruited from an OSA population, aged over 18. Participants will consist of male and female patients diagnosed with moderate-severe OSA (Apnea Hypopnea Index (AHI) greater than or equal to 15 per hour. Eligible participants, according to the protocol approved by the Northern X Region Ethics Committee, providing written informed consent will be enrolled into the study. Patients will be enrolled sequentially according to the randomisation list. Patients will be randomised to CPAP or SPAP.

The therapeutic pressure will be based on the most recent titration night of each patient. Comparisons between data will be made using a one-tailed t-test for non-inferiority of the SPAP algorithm compared with conventional CPAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years with mild-to-severe OSA (Apnea Hypopnea Index equal to or greater than 5 per hour).

Exclusion Criteria:

* Any medical condition which contraindicates (see Appendix A) the use of CPAP or AutoCPAP.
* Unstable cardiovascular disease (untreated or resistant hypertension acceptable).
* Unstable psychiatric disease.
* Other significant sleep disorder.
* Inability to tolerate CPAP due to nasal obstruction or claustrophobia, as determined by the investigation investigator.
* Any known factor or disease that might interfere with treatment compliance, investigation conduct or interpretation of the results such as psychiatric disease, history of non compliance to medical regimens, or unwillingness to comply with investigational requirements.
* Participation in another clinical trial in the previous month.
* Less than 2 hours recorded sleep in either arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
AHI | one post study night (once PSG is scored)
  The apnea hypopnea index (AHI) is a measure of sleep disordered breathing. It will be measured and compared between the two groups. The units are number of events per hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Fisher and Paykel Healthcare Sleep Lab, Auckland, New Zealand